CLINICAL TRIAL: NCT05463471
Title: Effect of Balanced Saline Solution and Albumin on Volume Expansion in Shock Patients: a Prospective Randomized Controlled Study
Brief Title: Effect of Balanced Saline Solution and Albumin on Volume Expansion in Shock Patients
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PUMCH-ICU-LY
Record Dates: First submitted 2022-06-20; First posted 2022-07-19 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Shock
Keywords: shock; sodium acetate ringer; albumin
MeSH Terms: conditions — Shock | interventions — Albumins

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sodium acetate ringer (Experimental)
  Interventions: Drug: Compound sodium acetate ringer injection
- albumin (Active Comparator)
  Interventions: Drug: Albumin

INTERVENTIONS:
Drug: Compound sodium acetate ringer injection — Quickly infuse 500ml of compound sodium acetate ringer injection for volume expansion within 20-30 minutes
  Arms: sodium acetate ringer
Drug: Albumin — Quickly infuse 500ml of albumin for volume expansion within 20-30 minutes
  Arms: albumin

SUMMARY:
To compare the direct effect of sodium acetate ringer injection or albumin on volume expansion in shock patients, and to provide reference for volume resuscitation strategy in shock patients

DETAILED DESCRIPTION:
CI/SVI increase amplitude and maintenance time

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old, gender unlimited
2. Shock requires volume resuscitation:

   Insufficient tissue perfusion: wet and cold skin, decreased urine volume (<0.5ml/kg/h), change of consciousness, blood lactate >2.0mmol/l or vasoactive drugs are required to maintain map>65mmhg
3. Presence of volume reactivity: (under controlled ventilation) PPV ≥ 15% or passive leg raising test (+) or (under controlled ventilation) IVC variability ≥ 18% or the presence of volume reactivity as judged by clinicians
4. The patient has no obvious restlessness, RASS ≤ 0
5. The legal representative of the subject signs the informed consent form-

Exclusion Criteria:

1. Pregnant and lactating women
2. End stage patients
3. BMI ≤ 15 or BMI ≥ 50
4. Contraindication of indwelling central vein catheter and invasive arterial catheter
5. Patients in ECMO and / or IABP therapy
6. Hemorrhagic shock, blood products such as concentrated red blood cells, plasma and platelets will be infused within 1 hour
7. Myocardial infarction, NYHA grade IV
8. Patients with hyperkalemia, hypercalcemia, hypermagnesemia and hypothyroidism
9. Allergic to compound sodium acetate ringer injection or albumin or with known side effects
10. Other factors that may affect the monitoring and evaluation of relevant indicators

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2025-12-12 (Estimated); Study Completion 2027-12-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of Cardiac output Index(CI) change | 2 hour
  The changes of cardiac output index before and after volume expansion were compared
Percentage of Stroke Volume Index（SVI）change | 2 hour
  The changes of Stroke Volume Index before and after volume expansion were compared

SECONDARY OUTCOMES:
Duration of Cardiac output Index(CI) change | 2 hour
  The duration of cardiac output index changes before and after volume expansion was compared
Duration of Stroke Volume Index（SVI）change | 2 hour
  The duration of Stroke Volume Index changes before and after volume expansion was compared

IPD SHARING:
Plan to Share IPD: No